CLINICAL TRIAL: NCT01691703
Title: Combined Technique Using Videolaryngoscopy and Bonfils for a Difficult Airway Intubation
Brief Title: Combined Technique for Difficult Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Barbe Pieters, MD, Catharina Ziekenhuis Eindhoven
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: COM.12; 12-624 (Other: Medisch Ethische Commissie Catharina Ziekenhuis Eindhoven)
Record Dates: First submitted 2012-09-18; First posted 2012-09-25 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Intubation; Difficult; Failed or Difficult Intubation; Failed or Difficult Intubation, Initial Encounter; Anesthesia Intubation Complication
Keywords: Fiber Optic Technology/methods; Intubation, Intratracheal/methods; Laryngoscopy/methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Videolaryngoscope and Bonfils (Experimental): First, the Macintosh videolaryngoscope (Karl Storz, Tuttlingen, Germany) will be used to achieve the best possible view and space of the laryngeal inlet for the insertion and manoeuvring of the Bonfils® (Karl Storz, Tuttlingen, Germany). Once the anaesthesiologist considers the view achieved to be the best view possible, a picture will be taken using C-CAMTM for C-MAC (Karl Storz, Tuttlingen, Germany), not showing any part of the videolaryngoscope. Thereafter the Bonfils® intubation scope, which will be preloaded with the endotracheal tube, will be brought into position in front of the laryngeal inlet. Again a picture not showing any part of one of the two devices will be taken. Once the Bonfils® has entered the trachea, the tracheal tube will be placed in the correct position.
  Interventions: Device: Videolaryngoscope and Bonfils

INTERVENTIONS:
Device: Videolaryngoscope and Bonfils — First, the Macintosh videolaryngoscope (Karl Storz, Tuttlingen, Germany) will be used to achieve the best possible view and space of the laryngeal inlet for the insertion and manoeuvring of the Bonfils® (Karl Storz, Tuttlingen, Germany). Once the anaesthesiologist considers the view achieved to be the best view possible, a picture will be taken using C-CAMTM for C-MAC (Karl Storz, Tuttlingen, Germany), not showing any part of the videolaryngoscope. Thereafter the Bonfils® intubation scope, which will be preloaded with the endotracheal tube, will be brought into position in front of the laryngeal inlet. Again a picture not showing any part of one of the two devices will be taken. Once the Bonfils® has entered the trachea, the tracheal tube will be placed in the correct position.
  Other Names: Macintosh videolaryngoscope (Karl Storz); Bonfils® (Karl Storz)

SUMMARY:
A difficult tracheal intubation can be a problem, even if one has taken all precautions. A possible solution can be using a videolaryngoscope in conjunct with the Bonfils® intubation scope. As such, the videolaryngoscope can be used to achieve the best possible view and space of the laryngeal inlet for the insertion and manoeuvring of the Bonfils® intubation scope.

DETAILED DESCRIPTION:
In this blinded, unrandomised trial the investigators would like to investigate the change in Cormack and Lehane grade when using both videolaryngoscope (Macintosh videolaryngoscope, Karl Storz, Tuttlingen, Germany) and Bonfils® (Karl Storz, Tuttlingen, Germany). They also want to record the success of intubation and the time needed until successful endotracheal intubation when using this technique as well as complications (trauma to the oral cavity, dental trauma, and regurgitation seen by the anaesthesiologist) that may occur. Also saturation (SpO2) at the end of the procedure will be noted and adjuncts that are used.

ELIGIBILITY:
Inclusion Criteria:

* Informed patient consent Age > 18 years History of difficult intubation (Cormack and Lehane III-IV)

One or more predictors of a difficult intubation:

* restricted neck movement
* thyromental distance < 60 mm
* interincisor/interdental distance < 30mm
* BMI > 35 kg.m-2 Elective surgery making endotracheal intubation necessary (other than head and/or neck surgery) Fasted (≥ 6 hours)

Exclusion Criteria:

* No informed patient consent Age < 18 years Emergency surgery, head and/or neck surgery Fasted < 6 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Cormack and Lehane grade achieved when using the combination technique compared with the Cormack and Lehane grade achieved earlier when using the Macintosh (video)laryngoscope alone. | The patients will be followed during induction of anesthesia, an average of 10 minutes
  The operator will score these grades during the process of intubation. Pictures will be taken of the first and the second Cormack and Lehane grade, and these pictures will later be scored by two anaesthesiologists, blinded for the technique used (videolaryngoscopy alone or videolaryngoscopy combined with the Bonfils®).

SECONDARY OUTCOMES:
Proportion of successful intubation with the 2 methods under study, without the use of adjuncts. | The patients will be followed during induction of anesthesia, an average of 10 minutes
  Proportion of successful intubation with the 2 methods under study, without the use of adjuncts.
Time until successful endotracheal intubation | The patients will be followed during induction of anesthesia, an average of maximal 3 minutes
  Time until successful endotracheal intubation will be defined as the time from the moment the blade of the Macintosh videolaryngoscope is placed between the teeth until the time the anaesthesiologist confirms the endotracheal tube to be in the trachea.
Complications rendered on during the procedure | The patients will be followed during induction of anesthesia, an average of 10 minutes
  Complications that will be recorded are: trauma to the oral cavity (defined as any amount of bright red blood in the oral cavity), dental trauma, and regurgitation seen by the anaesthesiologist. Also oxygen saturation (SpO2) at the end of the procedure will be noted, a saturation of less than 90% will be defined as hypoxia.
Adjuncts being used | The patients will be followed during induction of anesthesia, an average of 10 minutes
  Adjuncts that can be used are: gum elastic bougie, stylet and the BURP manoeuvre (performed by a second operator).

CONTACTS AND LOCATIONS:
Overall Officials: Barbe MA Pieters, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis Eindhoven, Eindhoven, Netherlands

REFERENCES:
- [Background] Van Zundert AA, Pieters BM. Combined technique using videolaryngoscopy and Bonfils for a difficult airway intubation. Br J Anaesth. 2012 Feb;108(2):327-8. doi: 10.1093/bja/aer471. No abstract available. PMID 22250284